CLINICAL TRIAL: NCT03793569
Title: Does Enhancing Maternal Peer Interactions Decrease Rates of Postpartum Depression?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Brittany Massare, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007890
Record Dates: First submitted 2018-06-05; First posted 2019-01-04 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Control group and intervention group. Intervention group will participate in peer discussion group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants will be recruited and asked to complete Edinburgh Postnatal Depression Scale (EPDS) at specific timepoints postpartum.
- Intervention group (Experimental): Participants will be recruited, asked to complete Edinburgh Postnatal Depression Scale at specific timepoints postpartum, and attend a peer discussion group.
  Interventions: Behavioral: Peer discussion group

INTERVENTIONS:
Behavioral: Peer discussion group — Subjects in the intervention group will be asked to attend one peer group between four and eight weeks postpartum. Peer groups will be expected to last approximately one hour. Each peer group will include 5-10 new mothers. A facilitator will be present for these groups, but the hope is to have mothers discuss with each other their postpartum experience and activities of their newborn at home.
  Arms: Intervention group

SUMMARY:
The long-term goal of this study is to validate a simple and inexpensive intervention to reduce the incidence and impact of Postpartum Depression (PPD). The central hypothesis is that enhancing social support of new mothers specifically via an organized peer get-together will decrease rates of postpartum depression. The rationale for the proposed research is that even though PPD is common and risk factors for developing PPD are known, simple and inexpensive interventions to prevent PPD need to be studied. Postpartum mothers will be recruited for the study and randomized into control versus intervention group. The intervention group will be placed in a peer discussion group. Incidence of PPD will be tracked.

DETAILED DESCRIPTION:
According to a 2014 Cochrane Review, postpartum depression (PPD) is present in 13% of new mothers by twelve weeks postpartum. Infant feeding, sleep routines, growth, and socioemotional and cognitive development can be adversely affected by maternal PPD. These negative effects can last into childhood. Previous studies have shown that strong social support is protective against PPD. The 2014 Cochrane Review on this topic comments that simple, inexpensive interventions to decrease rates of PPD are needed and that interventions led by lay-people and done in groups may be helpful to decrease rates of PPD. More recent studies focus on interventions for mothers already showing symptoms of postpartum depression, not on preventing these symptoms from developing.

The proposed work is important, because it capitalizes on recommendations for future research from the 2014 Cochrane Review on Psychosocial and Psychological Interventions for Preventing Postpartum Depression. The proposed work is also innovative, because it involves a preventive intervention from lay-people in a group setting, with new moms benefiting from each other. At the completion of this project, it is our expectation that mothers in the intervention group will have sustained decreased rates of PPD.

ELIGIBILITY:
Inclusion Criteria:

1. Women who deliver at the Hershey Medical Center
2. Postpartum women within first week after delivery
3. Women who are 18 years of age or older

Exclusion Criteria:

1. Postpartum women who delivered newborn before 35 0/7 gestational age.
2. Postpartum women whose newborn required any length of stay in the newborn intensive care unit.
3. Postpartum women who do not speak English.
4. Postpartum women who are less than 18 years old.
5. Postpartum women who are unable to provide consent.
6. Postpartum women who were on antidepressant or antianxiety medication or undergoing therapy for depression or anxiety during pregnancy or during postpartum hospitalization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Risk of development of postpartum depression | 4-8 weeks postpartum
  Edinburg Postnatal Depression Scale. Score 0-30. Score > or = 10 considered greater risk of depression.
Development of postpartum depression | 12 weeks postpartum
  Edinburg Postnatal Depression Scale. Score 0-30. Score > or = 10 considered greater risk of depression.
Development of postpartum depression | 6 months postpartum
  Edinburg Postnatal Depression Scale. Score 0-30. Score > or = 10 considered greater risk of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany A Massare, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No